CLINICAL TRIAL: NCT03406728
Title: Virtual Reality Can be Used to Improve Balance Reducing Dynamic Falls in Those With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDRC
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Virtual Reality; Training; Balance; Falls; PDSAFEX
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PDSAFEX GROUP (Active Comparator): Parkinson's Disease Sensory Attention Focused Exercise (PDSAFEX) is an exercise intervention developed in light of research which focuses on utilizing sensory integration and proprioception to improve balance. This intervention will be administered to one group of my participants. The protocol will be followed and led by trained volunteers.
  Interventions: Other: PDSAFEX
- CONTROL GROUP (Active Comparator): The control group in this study will be asked to maintain their daily lifestyle as closely as possible for the 12-week duration of the study.
  Interventions: Other: CONTROL
- VIRTUAL REALITY GROUP (Experimental): Virtual reality intervention will be assigned to this group. They will complete activities aimed at improving their dynamic balance. These activities are specifically developed based on previous literature and geared towards mirroring day to day activities/scenarios that individuals with PD may come into contact with.
  Interventions: Device: VIRTUAL REALITY

INTERVENTIONS:
Other: PDSAFEX — PDSAFEX is a week by week, progressive, exercise protocol that is followed. It lasts 12 weeks.
  Arms: PDSAFEX GROUP
Other: CONTROL — Participants will be asked to maintain their day to day life as consistently as possible for the 12 week duration of the study.
  Arms: CONTROL GROUP
Device: VIRTUAL REALITY — WorldViz Oculus Rift Move package (headset and software).
  Arms: VIRTUAL REALITY GROUP

SUMMARY:
This study aims to explore the use of full immersion virtual reality technology on improving balance in those with Parkinson's Disease. Patients will be immersed in a virtual environment and be tasked with completed games and activities, which mirror activities of daily living. It is hypothesized that this immersion in the virtual reality environment will improve their sensory pathways which are used to improve balance, decreasing falls.

DETAILED DESCRIPTION:
I will utilize a randomized independent measures single blind study. Meaning participants will be randomly assigned to three different groups. The randomization process will be completed by the primary investigator, using a computer randomization software. Essentially, participants will all be given numbers which will be entered into the software, which then randomly assigns them to one of the three groups. The groups are: the virtual reality intervention group, the PDSAFEX group and the control group. Dr. Almeida, the tester of UPDRS scores, will be unaware of which groups each participant is in - only I will be aware. I aim to recruit about thirty-six individuals (12 per group). The study will last twelve weeks. It will include: pre-testing and post-testing with a one month follow up. However, due to time constrains the post testing may be completed after 8 weeks so I can begin to analyze data and have a write up for my classmates and professors. There will still be the scheduled post testing and follow up after the fact at the specified original times (12 weeks and 1 month follow up). Participants will come into the MDRC three times per week. Depending on their group they will complete the PDSAFEX training or VR training intervention. PDSAFEX is a scripted intervention run by trained volunteers, it progresses in difficulty week by week. The VR technology group will complete a protocol that is associated with the software system of the device. They will be asked to complete exercises and/games aimed specifically at improving balance. For example, a game where they must dodge incoming objects while maintain good balance. Virtual reality, is also able to be increased in difficulty through changing the environment and/or stimuli characteristics/speed.

The virtual reality group will be exposed to the virtual reality simulation software for about 1 hour and 15 minutes including set up. They will complete a set of activities, games and exercises that are centered around improving balance. The activities and games are included in the software. The environment and difficulty of the protocol can be altered to make it more/less difficult depending on the participant's ability and/progression throughout the study.

The PDSAFEX intervention was created to improve an individual's sensory integration with a focus on improving balance. It consists of a 12-week protocol administered by trained volunteers. Each session lasts about 1 hour. Each week of the PDSAFEX protocol increases in either difficulty/volume to allow consistent improvements. Furthermore, some of the conditions/exercises are attempted under dim lights or with eyes closed to further stress the focus on limiting visual domains. Focusing on proprioception.

The control group will come in to the MDRC facility, to complete testing (pre, post and follow up). The participants in this group will be asked to continue their lifestyles without any drastic changes for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed with diagnosis with Parkinson's Disease by a registered movement disorders specialist
* Either gender
* Currently taking dopaminergic medication
* Able to walk 15m, unassisted
* Able to stand for 2 minutes unassisted
* Able to understand English Instructions
* Normal or corrected visions

Exclusion Criteria:

* Any other neurological disorder
* MoCa Score less than 18
* Commonly experiences vertigo, dizziness or motion sickness
* Seizures or dizziness due to light

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01-21 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  Assesses the burden and extent of Parkinson's Disease over the course of the disease.
Change in Sensory Organization Tests (SOT- 6) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  The sensory organization test is a set of six tests which measures an individuals balance under six different conditions. More specifically, it assess quantitative data about visual, proprioceptive and vestibular cues in order to maintain postural stability in stanceIt is completed using the Biodex machine.
Change in the number of Falls utilizing a Fall Calendar | The calendar will be completed daily but the results handed in at the end of each month for the duration of the study. The study will last three months, as such there should be three completed calendars.
  Subjective response that identifies the number of falls an individual participant has experienced. Participants will be supplied with a falls calendar which they will fill out and bring back in to the primary researcher.

SECONDARY OUTCOMES:
Change in Timed up and Go (TUG) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  The timed up and go test is an objective measure of balance, walking ability and fall risk in older adults.
Change in Activities Specific Balance Confidence scale (ABC scale) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  A subjective measure of confidence in completing certain activities of daily living or ambulatory actions without falling or experiencing unsteadiness.
Change in Gait Analysis | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  Measurement of an individuals step length, stride length, step variability and center of pressure. The results are all computed through the software; it provides you with all of the results after each trial of the test.
Change in Falls Efficacy Scale (FES) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  Assesses the perception of balance, stability and the fear of falling during activities of daily living.
Change in Parkinson's Disease Questionnaire (PDQ-39) | Pre test (a week prior), post test after 8 weeks and follow up with a washout period one month after completion of study.
  A self report questionnaire which assesses an individual's Parkinson's specific health quality over quality over the last month, their experience and difficulties in completing activities in the eight quality of life dimensions and the impact of Parkinson's on specific areas of wellbeing and functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Quincy J Almeida, PhD, Study Director — SunLife Movement Disorders Research and Rehabilitation Center
Locations (1):
- Sun Life Financial Movement Disorders Research and Rehabilitation Centre, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

DOCUMENTS (1):
  • Informed Consent Form (2018-01-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03406728/ICF_000.pdf